CLINICAL TRIAL: NCT03844828
Title: Clinical Study to Investigate Rotational Stability, Visual Performance, Contrast Sensitivity, Patient Satisfaction and PCO Rate After Implantation of a Trifocal Toric IOL
Brief Title: Clinical Study to Investigate Outcomes of Trifocal Toric IOL POD FT in Asian Eyes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY1901
Record Dates: First submitted 2019-02-13; First posted 2019-02-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cataract; Lens Opacities; Presbyopia
Keywords: Intraocular Lens; Trifocal; Toric Lens
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POD FT IOL Implantation experimental (Experimental): Mono- or bilateral implantation of trifocal toric intraocular lenses POD FT and POD F.
  Interventions: Device: IOL implantation experimental

INTERVENTIONS:
Device: IOL implantation experimental — Mono- or bilateral implantation of trifocal toric intraocular lenses POD FT. If both eyes of the same patient qualify for the implantation of a trifocal toric lens, a bilateral implantation will be performed. If only one eye qualifies for a trifocal toric lens, the contralateral eye will be implanted with the spherical trifocal IOL POD F (both lenses: (PhysIOL, Liège, Belgium).
  Other Names: POD FT IOL implantation

SUMMARY:
Prospective, controlled, single-surgeon, single-center clinical study to compare visual acuity outcomes to data obtained in a similar study by the same principal investigator on the trifocal IOL POD F (study no. PHY1802, ClinicalTrials.gov ID: NCT03688425)

DETAILED DESCRIPTION:
This is a prospective, controlled, single-surgeon, single-center clinical study, whereby patients undergoing routine cataract surgery will have mono- or bilateral implantation of trifocal toric intraocular lenses POD FT. The study is aimed to compare visual acuity outcomes the FineVision POD FT IOL to data obtained in a similar study by the same principal investigator on the trifocal FineVision POD F IOL (study no. PHY1802, ClinicalTrials.gov ID: NCT03688425), whereby patients undergoing routine cataract surgery will have bilateral implantation of trifocal intraocular lenses. The patients will either be implanted with the FineVision POD FT IOL in both eyes or, in case the corneal astigmatism in one of the two eyes of the same patient is too small to implant a toric lens, the FineVision POD F IOL will be implanted in this eye (both lenses: PhysIOL, Liège, Belgium).

The devices under investigation (FineVision POD FT and POD F) are trifocal glistening-free acrylic intraocular lenses (IOLs) manufactured by the sponsor of this study PhysIOL sa/nv. The main difference between the lenses is that that the POD FT IOL is the toric version of the POD F IOL. The IOLs will be implanted as part of the routine cataract surgery on patients suffering from cataract development.

Subjects participating in the trial will attend a total of 11 study visits (1 preoperative, 2 operative and 8 postoperative) over a period of 24 months. Subjects would have the option for unscheduled visits if required medically.

Primary endpoint data will be collected at the 6 months follow up visit and secondary endpoint data will be collected at the 1 Day, 1 Week, 1 month, 6, 12 and 24 months postoperative visits. Data analyses will be done after the last patient finished the final examination to support the study publication plan

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ages 45 years or older on the day of screening who have cataract(s) in one or both eyes or suffer from presbyopia;
* Regular corneal astigmatism ≥0.75 dioptres (measured by an automatic keratometer or biometer) in one or both eyes;
* Capability to understand and sign an IRB approved informed consent form and privacy authorization;
* Clear intraocular media other than cataract;
* Calculated IOL power is within the range of the study IOLs;
* Dilated pupil size large enough to visualize IOL axis markings postoperatively;
* Willing and able to conform to the study requirements.

Exclusion Criteria:

* Regular corneal astigmatism <0.75 dioptres (measured by an automatic keratometer or biometer) in both eyes
* Irregular astigmatism;
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal or optic disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse;
* Subjects with AMD suspicious eyes as determined by OCT examination;
* Subjects who may be expected to require retinal laser treatment during the course of the study or at a greater risk of developing cystoid macular edema;
* Previous intraocular or corneal surgery;
* Traumatic cataract;
* History or presence of macular edema;
* Pregnant, lactating or, if able to bear children, unwilling to use medically acceptable birth control over the course of the study;
* Concurrent or previous (within 30 days) participation in another drug or device investigation;
* Instability of keratometry or biometry measurements;
* Ocular hypertension or glaucoma;
* Significant dry eye;
* Unsuitable for study participation for any other reason, as determined by Investigator's clinical judgment (reason to be documented on eCRF).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2025-11-22 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Monocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions. | 6 months (120-180 days) postoperative
  Monocular visual acuity outcomes on CDVA under photopic light conditions are statistically non-inferior to data obtained in a similar study by the same principal investigator on the trifocal IOL POD F (study no. PHY1802, ClinicalTrials.gov ID: NCT03688425).

SECONDARY OUTCOMES:
Manifested refraction | Pre-OP, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2014. This data will also be used to calculate the manifested refractive spherical equivalent (MRSE)
Pupil Size | 6 months postoperative
  Photopic and mesopic pupil diameters are measured with a precision of at least +/-0.5 mm. For the photopic pupil diameters, eye illumination should be identical to that used for photopic contrast sensitivity testing. For the mesopic pupil diameters, eye illumination should be identical to that used for mesopic contrast sensitivity testing. It is required that pupil measurements be made with an infrared pupillometer / CCD camera. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 10 minutes).
  The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Uncorrected Distance Visual Acuity (UDVA) - monocular | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions.
Uncorrected Distance Visual Acuity (UDVA) - binocular | 6 months postoperative, 12 months postoperative, 24 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions.
Corrected Distance Visual Acuity (CDVA) - monocular | Pre-OP, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions.
Corrected Distance Visual Acuity (CDVA) - binocular | 6 months postoperative, 12 months postoperative, 24 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions.
Uncorrected Intermediate Visual Acuity at 70cm (UIVA) - monocular | 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  UIVA is measured with ETDRS charts placed in 70cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions.
Uncorrected Intermediate Visual Acuity at 70cm (UIVA) - binocular | 6 months postoperative, 12 months postoperative, 24 months postoperative
  UIVA is measured with ETDRS charts placed in 70cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions.
Distance Corrected Intermediate Visual Acuity at 70cm (DCIVA) - monocular | 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  DCIVA is measured with ETDRS charts placed in 70cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions.
Distance Corrected Intermediate Visual Acuity at 70cm (DCIVA) - binocular | 6 months postoperative, 12 months postoperative, 24 months postoperative
  DCIVA is measured with ETDRS charts placed in 70cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions.
Distance Corrected Intermediate Visual Acuity at 70cm (DCIVA) - monocular mesopic. | 6 months postoperative, 12 months postoperative, 24 months postoperative
  DCIVA is measured with ETDRS charts placed in 70cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under mesopic conditions.
Uncorrected Near Visual Acuity at 35cm (UNVA) - monocular | 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  UNVA is measured with ETDRS charts placed in 35cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions
Uncorrected Near Visual Acuity at 35cm (UNVA) - binocular | 6 months postoperative, 12 months postoperative, 24 months postoperative
  UNVA is measured with ETDRS charts placed in 35cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions
Distance Corrected Near Visual Acuity at 35cm (DCNVA) - monocular | 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  DCNVA is measured with ETDRS charts placed in 35cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions
Distance Corrected Near Visual Acuity at 35cm (DCNVA) - binocular | 6 months postoperative, 12 months postoperative, 24 months postoperative
  DCNVA is measured with ETDRS charts placed in 35cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions
Distance Corrected Near Visual Acuity at 35cm (DCNVA) - monocular mesopic | 6 months postoperative, 12 months postoperative, 24 months postoperative
  DCNVA is measured with ETDRS charts placed in 35cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under mesopic conditions
Defocus Curve | 6 months postoperative
  To assess the visual acuity for different distances, defocus curves under photopic light conditions are measured. This test is performed with best distance corrected refraction and spherical additions ranging from -5.0 D to +1.5 D. This examination is performed binocularly.
Binocular Contrast Sensitivity under photopic light conditions | 6 months postoperative, 12 months postoperative, 24 months postoperative
  Contrast Sensitivity under photopic light conditions using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Binocular Contrast Sensitivity under mesopic light conditions | 6 months postoperative, 12 months postoperative, 24 months postoperative
  Contrast Sensitivity under mesopic light conditions using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Binocular Contrast Sensitivity under mesopic light conditions and using a glare source | 6 months postoperative, 12 months postoperative, 24 months postoperative
  Contrast Sensitivity under mesopic light conditions with a glare source using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Patient reported outcomes | 6 months postoperative, 12 months postoperative
  Outcomes measures of a questionnaire to address the general patient satisfaction and possible side effects of the treatment. For this study, the validated and verified questionnaire Quality of Vision (QoV) und Near Activity Visual Questionnaire (NAVQ) will be used.
Slitlamp examination - Corneal Status | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Corneal Status
Fundus examination with dilated pupil | Pre-OP, 1 month postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Fundus
Slitlamp examination - Signs of inflammation | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  * Signs of inflammation
  * Anterior chamber cells,
  * Anterior chamber flare,
  * Cystoid macular oedema,
  * Hypopyon, and
  * Endophthalmitis
Slitlamp examination - Pupillary block | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Pupillary block
Slitlamp examination - Retinal detachment | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Retinal detachment
Slitlamp examination - Status of anterior and posterior capsule | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Status of anterior and posterior capsule
Slitlamp examination - IOL decentration | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL decentration
Slitlamp examination - IOL tilt | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL tilt
Slitlamp examination - IOL discoloration | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL discoloration
Slitlamp examination - IOL opacity | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL opacity
Photograph of IOL with dilated pupil to asses IOL rotation | OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  This examination shall only be performed in eyes implanted with POD FT lenses. To determine the rotational stability of the toric lenses after implantation, the actual IOL orientation has to be recorded as the intended surgical position during surgery using a photograph through the surgery microscope or other technique in order to document the rotational position of the IOL. Additional orientations are measured and recorded at the follow up visits by taking retroilluminated photographs in mydriasis using the slit lamp.
  To determine the rotational stability it is important that the IOL axis marks of the toric IOL are visible as well concurrent structures of the eye (in the same image) that are fixed and stable. Preferred fixed structures are limbal vessels. The pupil is dilated if necessary to visualize the IOL axis marks.

OTHER OUTCOMES:
Intraocular pressure (IOP) measurement | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The IOP will be measured with non-contact tonometer as part of the routine follow up examinations. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Keratometry | Pre-OP
  Keratometric measurements are performed to calculate the required IOL power. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Biometry | Pre-OP
  Biometry measurements are performed to calculate the required IOL power. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
IOL power and target refraction | Operative (day of Surgery)
  The parameter of the implanted IOL must be recorded as well as the target refraction given by the IOL calculator. This parameter is needed to calculate the accuracy of achieving the target refraction. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Fundus OCT | Pre-OP
  An OCT (optical coherence tomography) image will be taken at the preoperative visit to identify AMD suspicious eyes that need to be excluded from this study. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Edward Ang, MD, Principal Investigator — Asian Eye Institute
Locations (1):
- Asian Eye Institute, Makati City, Philippines

IPD SHARING:
Plan to Share IPD: No